CLINICAL TRIAL: NCT05758142
Title: Potassium Intake-response Trial to Control Hypertension
Acronym: PITCH
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The Principal Investigator moved to a new institution and funding for the study was discontinued.
Sponsor: Tulane University (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Joshua Bundy, Assistant Professor, Tulane University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2022-590; 2P20GM109036-06A1 (NIH)
Record Dates: First submitted 2023-02-24; First posted 2023-03-07 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Blood Pressure
MeSH Terms: interventions — Potassium Chloride; Potassium, Dietary

STUDY DESIGN:
Intervention Model Description: Eligible participants will be randomly assigned to placebo or 1 of 3 active intervention groups in a 1:1:1:1 ratio.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The proposed trial will employ placebo control and blinding of participants and study staff recording participant information. A Bioinformatics and Biostatistics Core will control the randomization and intervention allocation, preserving the blinding of the investigators and study staff in charge of day-to-day operations. Study participants will receive potassium tablets or placebo and will be unaware of their placebo or dosing assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Placebo (Placebo Comparator): Participants randomized to the placebo arm will receive 1, 2, or 3 inert placebo tablets twice daily (i.e., 2, 4, or 6 tablets per day) for 12 weeks.
  Interventions: Other: Placebo
- Potassium Chloride 30 mmol per day (Active Comparator): Participants randomized to the 30 mmol per day group will receive 1 potassium chloride tablet (15 mmol strength) twice daily (i.e., 2 tablets per day) for 12 weeks.
  Interventions: Dietary Supplement: Potassium Chloride
- Potassium Chloride 60 mmol per day (Active Comparator): Participants randomized to the 60 mmol per day group will receive 2 potassium chloride tablets (15 mmol strength) twice daily (i.e., 4 tablets per day) for 12 weeks.
  Interventions: Dietary Supplement: Potassium Chloride
- Potassium Chloride 90 mmol per day (Active Comparator): Participants randomized to the 90 mmol per day group will receive 3 potassium chloride tablets (15 mmol strength) twice daily (i.e., 6 tablets per day) for 12 weeks.
  Interventions: Dietary Supplement: Potassium Chloride

INTERVENTIONS:
Dietary Supplement: Potassium Chloride — Oral administration of potassium chloride tablets
  Other Names: Klor-Con
  Arms: Potassium Chloride 30 mmol per day; Potassium Chloride 60 mmol per day; Potassium Chloride 90 mmol per day
Other: Placebo — Oral administration of inert placebo tablets
  Other Names: Zeebo
  Arms: Placebo

SUMMARY:
The Potassium Intake-response Trial to Control Hypertension (PITCH) will test the intake-response relationship between potassium supplementation and blood pressure, which may inform clinical guidelines on the optimal level of potassium supplementation for blood pressure lowering among adults with elevated blood pressure or hypertension and dietary guidelines for population intake.

DETAILED DESCRIPTION:
Hypertension is the leading preventable risk factor for cardiovascular disease (CVD) and all-cause mortality, and prevention and treatment of high blood pressure (BP) is crucial for reducing the global burden of CVD.

Nonpharmacological interventions, including dietary interventions, are recommended as the primary approach for prevention and treatment of elevated BP and hypertension in US adults. Observational epidemiological studies have reported an inverse association between dietary potassium intake and BP, and clinical trials have documented that potassium supplementation reduces BP. However, previous clinical trials of potassium supplementation and BP have been limited to comparing one single dose of potassium supplementation (mostly 60 mmol/day or 1173 mg/day) to placebo control. Therefore, the optimal level of dietary intake of potassium in the population is currently unknown. In 2019, the National Academies of Science, Engineering, and Medicine updated the Dietary Reference Intake (DRI) recommendations for potassium intake based on the most current evidence associating potassium intake with CVD outcomes, including BP. Limited evidence precluded the DRI Committee from establishing a Chronic Disease Risk Reduction Intake level. The specific goal of the proposed randomized controlled trial is to study the intake-response effect for 4 levels of potassium supplementation on BP among adults with elevated BP or hypertension (defined as average untreated office systolic BP 120-159 mm Hg and diastolic BP <100 mm Hg). The investigators will test the primary hypothesis that compared with placebo (0 mmol/day potassium supplementation), there is a progressive relationship between increasing doses of oral potassium supplementation (30, 60, and 90 mmol/day or 1173, 2346, 3519 mg/day) and decreasing levels of 24-hour systolic BP from baseline to 12-weeks of follow-up. The investigators will also evaluate effects on daytime (awake) and nighttime (asleep) BP, office systolic and diastolic BP, sodium excretion, and effect mediation and moderation by age, sex, race, central adiposity, baseline urine excretion of sodium and potassium, and change in urine sodium. The results from the proposed trial will fill a critical knowledge gap and may identify the optimal level of potassium supplementation for BP lowering among adults with elevated BP and hypertension. This information can be used to develop dietary guidelines for the prevention and treatment of elevated BP, hypertension, and CVD.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged >18 years of any race/ethnicity
* Elevated BP or hypertension at screening (untreated office systolic BP 120-159 and diastolic BP <100 mm Hg)
* Willing and able to provide informed consent

Exclusion Criteria:

* Medical condition in which potassium supplementation is contraindicated: history of heart failure, myocardial infarction, stroke, cardiac arrythmia, chronic kidney disease or estimated glomerular filtration rate <60 ml/min/1.73 m^2, diabetes or non-fasting glucose >200 mg/dL, major depressive disorder (PHQ-9 score ≥15), psychosis, ulcer diseases including esophageal-gastric ulcer, malignancy in the past 5 years, liver disease, organ transplant, Addison's disease (adrenal insufficiency)
* Use of medications which may alter serum potassium levels or in which potassium supplementation is contraindicated: antihypertensive agents, antihistamines, antiparkinson agents, antimuscarinic agents, antipsychotics, muscle relaxants, systemic corticosteroids, or chronic use of non-steroidal anti-inflammatory drugs
* Serum potassium ≥5.0 mEq/L
* Metabolic acidosis
* Consumption of >85th percentile of usual potassium intake among US adults (>3,750 mg/day)
* For women, current pregnancy, breastfeeding, or plans to become pregnant during the study
* Consumption of ≥21 alcoholic beverages per week or consumption of ≥6 beverages per occasion
* Current or planned residence making it difficult to meet trial requirements or travel to the study site
* Current participation in another intervention or pharmaceutical trial
* Unable or unwilling to complete 24-hour BP or urinary sample collection
* Other concerns regarding ability to meet trial requirements, at the discretion of the investigators or staff

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2023-03-29 (Actual); Primary Completion 2024-05-03 (Actual); Study Completion 2024-05-03 (Actual)

PRIMARY OUTCOMES:
Change in 24-hour systolic blood pressure (BP) from baseline to 12 weeks | 12 weeks
  Ambulatory blood pressure monitoring will be used to determine 24-hour systolic BP

SECONDARY OUTCOMES:
Change in 24-hour diastolic blood pressure (BP) from baseline to 12 weeks | 12 weeks
  Ambulatory blood pressure monitoring will be used to determine 24-hour diastolic BP
Change in daytime (awake) systolic blood pressure (BP) from baseline to 12 weeks | 12 weeks
  Ambulatory blood pressure monitoring will be used to determine daytime BP
Change in daytime (awake) diastolic blood pressure (BP) from baseline to 12 weeks | 12 weeks
  Ambulatory blood pressure monitoring will be used to determine daytime BP
Change in nighttime (asleep) systolic blood pressure (BP) from baseline to 12 weeks | 12 weeks
  Ambulatory blood pressure monitoring will be used to determine nighttime BP
Change in nighttime (asleep) diastolic blood pressure (BP) from baseline to 12 weeks | 12 weeks
  Ambulatory blood pressure monitoring will be used to determine nighttime BP
Change in office systolic blood pressure (BP) from baseline to 12 weeks | 12 weeks
  An automated oscillometric device will be used to determine office BP based on the mean of 6 blood pressure values from two 12-week visits minus the mean of 6 values from 2 baseline visits
Change in office diastolic blood pressure (BP) from baseline to 12 weeks | 12 weeks
  An automated oscillometric device will be used to determine office BP based on the mean of 6 blood pressure values from two 12-week visits minus the mean of 6 values from 2 baseline visits

CONTACTS AND LOCATIONS:
Overall Officials: Joshua D Bundy, PhD, MPH, Principal Investigator — Assistant Professor
Locations (1):
- Tulane University Office of Health Research, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Yes
The study data sharing plan will comply with all NIH policies for data sharing. Data sharing will be executed through the centralized NIH data repository and will be implemented in a timely manner. The study data, including data from baseline and follow-up visits, will be prepared for transmission to the NHLBI data repository - the Biologic Specimen and Data Repository Information Coordinating Center (BioLINCC). Data will be prepared by the study coordinating center and sent to the PO for review prior to release. These data will be free of identifiers that allow identification of individual research participants either directly or through "deductive disclosure." In addition, the investigators will offer, through a public access website, opportunities for outside investigators to collaborate using complete study data.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data sets will be submitted to the NIH Program Official (PO) no later than 3 years after the end of the final patient follow-up or 2 years after the main paper of the trial has been published, whichever comes first.
Access Criteria: Upon request